CLINICAL TRIAL: NCT05684133
Title: REMISE Study: REMnant Biospecimen Investigation in SEpsis
Acronym: REMISE
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Vanderbilt University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Christopher Seymour, Associate Professor, Dept. of Critical Care Medicine, University of Pittsburgh School of Medicine Associate Professor, Depts. of Emergency Medicine & Clinical Translational Science The CRISMA Center, Director, Translational and Clinical Science Program, University of Pittsburgh
Other Study IDs: STUDY21120013; 5R21GM144851-02 (NIH)
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Remnant/leftover blood samples collected after usual patient care in comparison to newly obtained blood samples to evaluate 1) validity and stability of remnant blood samples vs fresh, newly obtained blood samples. 2) blood proteins, biomarkers, and other -omics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sepsis: Adult patients (18 years or older) meeting Sepsis-3 criteria within 6 hours of emergency department admission. Patients will be excluded with the following conditions: traumatic injury, cardiac arrest, stroke, comfort measures only.

SUMMARY:
In the REMISE is study, we will compare blood proteins, biomarkers, and other -omics prospectively collected from patients with sepsis from two sources, i.) remnant (discarded) samples from the clinical laboratory, and ii.) prospectively collected in UPMC Presbyterian hospital research coordinator specimen collected biospecimens.

Analyses will include traditional biomarkers, quantitative proteomics, metabolomics, lipidomics, transcriptomics, and pathogen genomic sequencing in both sets of samples. This data will allow the assessment of the feasibility, integrity, and scientific value of remnant samples compared to research coordinator samples collected at the bedside for mechanistic sepsis research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, at least 18 years of age
* Meeting Sepsis-3 criteria within 6 hours of admission
* Biospecimens obtained for routine clinical care and measurement
* Peripheral intravenous access

Exclusion Criteria:

* Patients who do not have Sepsis-3
* Traumatic injury,
* Inability to consent or contact legal representative,
* Cardiac arrest,
* Stroke,
* Comfort measures only,
* Unable to obtain intravenous access, and/or
* Subject declines to participate.
* No residual blood left in clinical sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Sepsis-3 presenting to eligible emergency departments.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in traditional biomarkers, proteomics, pathogen sequencing, and metabolomics/lipidomics between prospectively collected biospecimens and remnant biospecimens. | 01/2024

SECONDARY OUTCOMES:
Measurement of traditional biomarkers in all samples | 1/2024
  Traditional biomarkers to be measured in remnant and research specimens including inflammatory and endothelial-related biomarkers.
Measurement of proteomics in all samples | 1/2024
  Proteomics to be measured in remnant and research specimens to capture over 50 different plasma proteins.
Measurement of metabolomics/lipidomics in all samples | 1/2024
  Metabolomics and lipidomics to be measured in remnant and research specimens to capture organic acids, amino acids, and phospholipids.
Pathogen sequencing in all samples | 1/2024
  Pathogen sequencing will be performed on all remnant and research specimens to precisely identify the causative strain(s) in the infection.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Seymour, M.D., Principal Investigator — University of Pittsburgh / UPMC
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided